CLINICAL TRIAL: NCT06577233
Title: Superior Hypogastric Nerve Plexus Block With Bupivacaine for Postoperative Pain Reduction Following Robotic Assisted Resection of Endometriosis: A Randomized Control Trial
Brief Title: Superior Hypogastric Nerve Plexus Block With Bupivacaine After Robotic Resection of Endometriosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, XIAOMING GUAN, Division Chief of Minimally Invasive Gynecologic Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-55139
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis
Keywords: Endometriosis, Postoperative Pain, Robotic Surgery
MeSH Terms: conditions — Endometriosis; Pain, Postoperative | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study will be a randomized single blind clinical trial where the participant will be blinded to whether they received a superior hypogastric nerve block with 0.25% Bupivacaine Hydrochloride (investigative treatment) or 0.9% normal saline (placebo). The researcher will not be blinded and will know which arm the participant has been randomized to. Randomization will be performed by a computer generator in RedCap.
Who Masked: Participant
Masking Description: The subject will be told that the study is regarding postoperative pain control and superior hypogastric nerve plexus blocks with bupivacaine hydrochloride and that they will be randomized into the placebo group or the intervention group, but will be blinded to their assignment. They will be informed they have a 50% chance of being randomized to the investigative treatment group and a 50% chance of being chance of being randomized to the placebo group. Risks and benefits of the procedure as well as consent for the procedure will be obtained. The subject will be assigned a number to de-identify the data and then be randomized using a computer generator and RedCap. The practitioner will be aware of the group that is assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigative Treatment (Experimental): During the surgery, the investigative treatment group will have 5cc of diluted 0.25% Bupivacaine Hydrochloride injected into the superficial retroperitoneal area over the superior hypogastric nerve plexus.
  Interventions: Drug: Bupivacaine Hydrochloride
- Placebo (Placebo Comparator): During the surgery, the placebo group will have 5cc of 0.9% normal saline injected into the superficial retroperitoneal area over the superior hypogastric nerve plexus.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — 10cc of 0.25% Bupivacaine Hydrochloride will be injected into the peritoneum overlying the superior hypogastric nerve plexus with a laparoscopic needle during robotic surgery
  Other Names: Marcaine
  Arms: Investigative Treatment
Drug: Normal saline — 10cc of 0.9% normal saline will be injected into the peritoneum overlying the superior hypogastric nerve plexus with a laparoscopic needle during robotic surgery
  Other Names: 0.9% Normal Saline
  Arms: Placebo

SUMMARY:
Endometriosis is a condition that causes significant pelvic pain and affects 10-15% of reproductive age women. Treatment options area both medical and surgical for pain relief, however with surgical options, past studies have demonstrated a higher risk of surgical complications as well as higher postoperative pain scores in women with endometriosis. Despite attempts to limit narcotic pain medications with enhanced recovery after surgery (ERAS) protocols, persistent opioid use after surgery is a national crisis, and it is important to explore multimodal options for pain relief. Various studies have shown improvement in pain with use of superior hypogastric nerve blocks in gynecologic surgery, but these effects have not yet been examined in the setting of a minimally invasive endometriosis resection.

The goal of this clinical trial is to determine if a superior hypogastric nerve plexus block with 0.25% bupivacaine hydrochloride can decrease postoperative pain and opioid requirements in patients undergoing robotic assisted resection of endometriosis for the first week after surgery.

Researchers will perform a superior hypogastric nerve plexus block by either injecting 0.25% bupivacaine hydrochloride (investigative treatment) or normal saline (placebo) in subjects who are undergoing a robotic assisted resection of endometriosis.

To determine if postoperative pain is reduced, the subject will be asked to rate their pain score on the Visual Analog Scale (VAS) at 0 hours, 2 hours and 4 hours postop while in the Post-anesthesia Care Unit (PACU). They will then document their pain score each day on a form provided to them for 7 days after surgery.

To determine the effect of this research study on postoperative opioid requirements, the subject will be asked to fill out a form documenting how many tablets of an opioid medication they took each day for a total of 7 days after surgery.

DETAILED DESCRIPTION:
This clinical study will recruit patients at their preoperative visit. If the surgery is Davinci single incision laparoscopic surgery (or single incision plus one port) for resection endometriosis, the subject will be informed about the clinical trial, as well as risks and benefits of enrolling by the fellow or attending surgeon. The pre-op visit is typically 1-4 weeks before the day of surgery. They can make the decision either the day of the pre-op visit or they can have time to consider it and inform us of their decision on the day of surgery. If they agree to participate in the trial, they will be consented for the procedure and for enrollment in the trial. The subjects that agree will be assigned a number to de-identify data and then randomly assigned to the placebo or interventional treatment group with use of a computer generator (RedCap). The clinician will be aware of the group that they are in but the subject will not be aware of the group assignment.

At the time of enrollment the subject will also be informed that their medical record will be accessed to obtain information from the surgery and demographics. They will be informed that this information will be de-identified and entered into a password protected database called RedCap. The subject information obtained that will be demographics including those obtained from their pre-operative visit clinic note such as: age, race and ethnicity, gravidity/parity, surgical history, preoperative visual analog scale (VAS) score. As well as the information obtained from the operative note: stage of endometriosis diagnosed, additional laparoscopic procedures performed during the surgery, operative time, estimated blood loss, major intraoperative complication, uterine weight, and pathology. Their medical records will be reviewed by members of the surgical team at the time of surgery, at their postoperative visit, and during data analysis, so three times total.

During the case, The trocar used for the robotic single site surgery is the Single-Site port with curved cannulas made for the DaVinci XI single site instruments. This is inserted through one incision in the umbilicus. If the patient has severe endometriosis, a right lower quadrant 8mm trocar is inserted. This is standard of care for robotic assisted single site resection of endometriosis.

For the block portion of the study, the placebo group will have 5cc of 0.9% normal saline injected superficially into the retroperitoneal space overlying the superior hypogastric nerve plexus just distal to the common iliac bifurcation, bilaterally (10cc normal saline total). The nerve plexus bifurcation will be identified by the sacral promontory and the injection region will be approximately 1-2cm below this area bilaterally. The interventional treatment group will have 5cc total of diluted 0.25% bupivacaine hydrochloride injected at the same location (10cc total).

We will perform the superior hypogastric nerve block with 10cc of 0.25% Bupivacaine Hydrochloride as this is the most common analgesic used for this block. Bupivacaine Hydrochloride is FDA approved for subcutaneous nerve blocks at concentrations of 0.25% and 0.50%. The Texas Children's Hospital Pharmacy is familiar with 0.25% Bupivacaine Hydrochloride as it is a commonly used medication in the operating room and is already present in the endometriosis resection set as it is typically injected in the incision sites after the surgery. The subject will be blinded to the group they are randomized to (either placebo or investigative treatment), but the operating room nurses and physicians will not be blinded. The surgical team will look at what group the subject is assigned to before the case and either ask for the nurse to get the 0.25% Bupivacaine Hydrochloride or a saline filled 10cc syringe. If they are In the 0.25% Bupivacaine Hydrochloride group, no additional medication will be ordered as it is already in the set.

With current endometriosis resection surgeries, 0.25% bupivacaine hydrochloride is used as local anesthetic at skin incisions and is part of the standard surgery bundle. The nerve block will be performed with instruments already in the surgery set and this will not be billed as a separate procedure. Thus, this block and the bupivacaine hydrochloride will not be expected to add to the cost of the surgery and the subject will not be charged.

The standard of care for endometriosis resection surgeries is no nerve block and to send the patient home with Ibuprofen, Tylenol and Oxycodone. The investigational treatment in this study will be to perform the nerve block, they will still go home with the same pain medications of Ibuprofen, Tylenol and Oxycodone with the same amount of pills prescribed.

To keep data safe and subject information protected, any physical data will be stored in a locked cabinet in the PI's office in Pavilion for Women. Subjects will be assigned numbers as participants so that all data can be de-identified. Electronic data will be kept in an online, password protected database (RedCap), This information will be de-identified and stored in Red-Cap, a web-based database that is password protected. As the information being put into Red-Cap will be de-identified, the information will be unable to be traced through the database. This will be secure as only the direct members of the research team will have access to this information. Red-Cap is a database that is useful to research studies as information does not need to be downloaded to specific computers or stored on external hard drives. By insuring the patient information is de-identified and untraceable before entering it into RedCap, it helps keep the data in one place password protected, therefore reducing the risks associated with losing external hard drives or personal computers.

The sample size was calculated by a Baylor College of Medicine Statistician. The proposed sample size will include 60 subjects from Texas Children's Hospital, with 30 subjects randomized to each arm. This was calculated to detect a 38% decrease in the proportion of subjects with VAS scores > 4 in the 2 hours post-op at the 95% confidence level with a power of 80%, which would come out to 25 subjects per group for a total of 50 subjects. We plan to add 20% to account for drop out rate, for a final number of 60 subjects (30 per group).

For statistical analysis, primary analysis includes comparing the Visual Analog Scale (VAS) pain levels at 2 hours, 4 hours and daily for 1 week after surgery between the placebo and the treatment group. This would be a comparison of means (mean VAS pain level score at each time in the placebo vs treatment group).

Secondary analysis includes calculating the amount of narcotic pain medications used in the first 24 hours and first week after surgery in morphine milligram equivalents and comparing that number between the placebo and treatment group. This would be a comparison of means (mean amount of narcotic pain medications in morphine milligram equivalents in the placebo vs treatment groups).

In order to reduce missing data or the subject not filling out the form, the Fellow surgeon will call the subject 7 days after surgery with a reminder to complete the form. If they do not do this, they will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Scheduled to undergo a robotic assisted resection of endometriosis

Exclusion Criteria:

* Subjects who are part of a vulnerable population will be excluded including those who are prisoners, younger than 18 years old, pregnant, individuals with mental disabilities or cognitive impairment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Postoperative pain level documented at 0, 2 and 4 hours after surgery, then once a day for 7 days after surgery.
  Postoperative pain levels as characterized by the Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Opioid use | The first 7 days after surgery
  The amount of opioid medication used in the immediate postoperative period in morphine milligram equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Guan, PhD, MD, Principal Investigator — Department Chair of Minimally Invasive Gynecologic Surgery
Locations (1):
- Texas Childrens Hospital Pavilion for Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zakim D, Herman RH. The effect of intravenous fructose and glucose on the hepatic alpha-glycerophosphate concentration in the rat. Biochim Biophys Acta. 1968 Oct 15;165(3):374-9. doi: 10.1016/0304-4165(68)90215-8. No abstract available. PMID 5737931
- [Background] Brunes M, Johannesson U, Habel H, Forsgren C, Moawad G, Ek M. Peri- and postoperative outcomes in patients with endometriosis undergoing hysterectomy. Eur J Obstet Gynecol Reprod Biol. 2022 May;272:104-109. doi: 10.1016/j.ejogrb.2022.02.180. Epub 2022 Mar 9. PMID 35299012
- [Background] Kanellos P, Nirgianakis K, Siegenthaler F, Vetter C, Mueller MD, Imboden S. Postoperative Pain Is Driven by Preoperative Pain, Not by Endometriosis. J Clin Med. 2021 Oct 15;10(20):4727. doi: 10.3390/jcm10204727. PMID 34682850
- [Background] Meyer LA, Lasala J, Iniesta MD, Nick AM, Munsell MF, Shi Q, Wang XS, Cain KE, Lu KH, Ramirez PT. Effect of an Enhanced Recovery After Surgery Program on Opioid Use and Patient-Reported Outcomes. Obstet Gynecol. 2018 Aug;132(2):281-290. doi: 10.1097/AOG.0000000000002735. PMID 29995737
- [Background] Aytuluk HG, Kale A, Astepe BS, Basol G, Balci C, Colak T. Superior Hypogastric Plexus Blocks for Postoperative Pain Management in Abdominal Hysterectomies. Clin J Pain. 2020 Jan;36(1):41-46. doi: 10.1097/AJP.0000000000000767. PMID 31567396
- [Background] De Silva P, Daniels S, Bukhari ME, Choi S, Liew A, Rosen DMB, Conrad D, Cario GM, Chou D. Superior Hypogastric Plexus Nerve Block in Minimally Invasive Gynecology: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2022 Jan;29(1):94-102. doi: 10.1016/j.jmig.2021.06.017. Epub 2021 Jun 29. PMID 34197956